CLINICAL TRIAL: NCT01897324
Title: Which is the Best IVF/ICSI Protocol to be Used in Poor Responders Receiving Growth Hormone as an Adjuvant Treatment ? A Prospective Randomized Study
Brief Title: IVF/ICSI Protocols in Poor Responders With Growth Hormone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, lecturer of obstetrics and gynecology, cairo university, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WHC2013
Record Dates: First submitted 2013-07-02; First posted 2013-07-11 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Female Infertility Due to Diminished Ovarian Reserve
Keywords: Poor Ovarian Response; Poor Responders; IVF/ICSI; Growth Hormone
MeSH Terms: interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- The Long protocol (Experimental): Patients in the group A received a long protocol of pituitary down-regulation with triptorelin (Decapeptyl; Ferring, Switzerland) which started on day 21 of preceding cycle at a dose of 0.1 mg/day. On the second day of menstruation HMG was started and this was associated with reduction of triptorelin to 0.05 mg/day. This reduced daily dose was administered until the day hCG was given. Growth hormone co-treatment was administrated on day 6 of HMG stimulation daily in a dose of 2.5 mg S.C. till the day of hCG administration.
  Interventions: Drug: Growth hormone (Norditropin, Novo nordisk)
- The Short protocol (Experimental): The short agonist protocol was started on cycle day 1 with triptorelin (Decapeptyl Ferring Pharmaceuticals, Germany) 0.05 mg/day S.C. Human menopausal gonadotropin IM daily (HMG 75 IU, Merional, IBSA) were also administered starting from days 2 to 3 of cycle. The dose was adjusted for each patient according to the diameter of the follicles detected in their follow up ultrasound. Growth hormone (Norditropin, Novo nordisk) was administrated on day 6 of HMG stimulation daily in a dose of 2.5 mg S.C. till the day of hCG administration.
  Interventions: Drug: Growth hormone (Norditropin, Novo nordisk)
- The Antagonist protocol (Experimental): Gonadotrophins IM daily (HMG 75 IU, Merional, IBSA)was administrated from day 2 of the cycle. Growth hormone (Norditropin, Novo nordisk) was administrated on day 6 of HMG stimulation daily in a dose of 2.5 mg S.C. till the day of hCG administration. The GnRH antagonist (Cetrotide) was given when the leading follicle was from 12 to 14 mm, at a daily dose of 0.25 mg SC.
  Interventions: Drug: Growth hormone (Norditropin, Novo nordisk)
- The Microflare protocol (Experimental): the patients in this group were given oral contraceptive pills (OCPs) for 28 days, this was followed by 2 days free. Triptorelin (Decapeptyl Ferring Pharmaceuticals, Germany) 0.05 mg/day S.C. was then started daily followed by human menopausal gonadotropin IM daily (HMG 75 IU, Merional, IBSA) 3 days later. Growth hormone (Norditropin, Novo nordisk) was administrated on day 6 of HMG stimulation daily in a dose of 2.5 mg S.C. till the day of hCG administration.
  Interventions: Drug: Growth hormone (Norditropin, Novo nordisk)

INTERVENTIONS:
Drug: Growth hormone (Norditropin, Novo nordisk)

SUMMARY:
in this study, we are trying to monitor the effect of the addition of growth hormone on the different down regulation protocols ( long, short, antagonist and microflare). The outcome will be primarily assessed by the clinical pregnancy rates.

DETAILED DESCRIPTION:
Poor responders undergoing IVF/ICSI cycles have emerged as a major problem. the need to find a proper stimulation protocol is a must. in this study we are trying to detect the best stimulation protocol ,in addition to growth hormone ,that can give the highest pregnancy rates in these patients.

ELIGIBILITY:
Inclusion Criteria:

ESHRE consensus 2011,At least two of the following three features must be present:

* Advanced maternal age (≥40 years) or any other risk factor for POR;
* A previous POR (≤3 oocytes with a conventional stimulation protocol);
* An abnormal ovarian reserve test (i.e. AFC < 5-7 follicles or AMH < 0.5 -1.1 ng/ml).

Exclusion Criteria:

* female patients with causes of infertility other than poor ovarian reserve
* females suffering from congenital or acquired uterine anomalies
* females with focal uterine lesions
* females who had previous ovarian surgeries
* females with history of previous exposure to radiotherapy , or chemotherapy
* females refusing to get enrolled in the study

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 287 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Numbers of oocytes retrieved and number of fertilized oocytes | 2 years
  Number of oocytes retrieved on the day of vaginal egg collection guided by trans vaginal ultrasound scan , 35 hours after hCG administration.

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- private IVF medical center, Giza, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Dakhly DM, Bayoumi YA, Gad Allah SH. Which is the best IVF/ICSI protocol to be used in poor responders receiving growth hormone as an adjuvant treatment? A prospective randomized trial. Gynecol Endocrinol. 2016;32(2):116-9. doi: 10.3109/09513590.2015.1092136. Epub 2015 Sep 29. PMID 26416521